CLINICAL TRIAL: NCT04742322
Title: Efficacy of Using Bifidobacterium Lactis CCT 7858 in Improving Gastrointestinal Symptoms in Adults Using Antibiotics
Brief Title: Efficacy of Bifidobacterium Lactis CCT 7858 in Adults Using Antibiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, Clinical Professor, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 40641120900005364
Record Dates: First submitted 2021-01-21; First posted 2021-02-08 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Surgery; Infection
Keywords: probiotic; antibiotic; B lactis
MeSH Terms: conditions — Infections | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1x capsule/day - maltodextrin, period of 10 to 14 days
  Interventions: Dietary Supplement: Maltodextrin
- B Lactis (Experimental): 1x capsule/day - 9x10x10 UFC, period of 10 to 14 days
  Interventions: Dietary Supplement: Bifidobacterium Lactis CCT7858

INTERVENTIONS:
Dietary Supplement: Bifidobacterium Lactis CCT7858 — Probiotic B Lactis
  Arms: B Lactis
Dietary Supplement: Maltodextrin — Maltodextrin
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of the probiotic Bifidobacterium lactis CCT 7858 in preventing and / or improving gastrointestinal symptoms in adults using antibiotics. For this, a randomized, double-blind, placebo-controlled clinical trial will be carried out. The sample will be composed of adults who will be recruited in a hospital, who have been hospitalized and receive a prescription for antibiotics. The individuals will be separated into two groups: intervention and placebo. 104 patients will be included, 52 for each group. Inclusion criteria:

adults of both sexes and aged between 18 and 65 years, who have been recruited within 24 hours after starting antibiotic treatment, the prescribed treatment should be with antibiotics for a minimum of 9 days and a maximum of 14 days. The informed consent must be signed before starting the study.

DETAILED DESCRIPTION:
Two groups (placebo and intervention) will receive supplementation, the Placebo group will receive maltodextrin and Intervention group will receive probiotic B. lactis, that should be consumed for a period of 10 to 14 days depending on the duration of administration of the antibiotic (should be consumed until 7 day after the last antibiotic).

As a way of ensuring an equal distribution of the number of participants in the study groups and ensuring that the groups are similar, a randomization by blocks will be carried out and stratified by sex and age. The program that will be used to generate random numbers is the Research Randomizer Form v4.0. The packaging of both supplements will be identical except for the color, which will distinguish maltodextrin from probiotic.

Supplements will be delivered by a research collaborator as a way to guarantee blinding.

The probiotic to be supplied will be Bifidobacterium lactis CCT 7858 (GABBIA® Biotechnology and Development, Santa Catarina, Brazil). The probiotic will be offered in capsule and in the concentration of 9x10 10 UFC.

The groups will be evaluated in two moments: baseline and final.

The evaluation of the individuals will be performed through the collection of the following data: necessity and duration of antibiotic therapy (type of antibiotic) used while participating in the study.

Blood pressure will also be assessed.

Body weight will be measured. The body mass index will be calculated

In order to verify the tolerance and effectiveness of the supplements, questions regarding the frequency and consistency of feces will be asked, evaluated using the Bristol scale (1: separate pieces, 2: segmented sausage shape, 3: cracked sausage shape, 4: smooth and soft sausage shape, 5: soft pieces, 6: aerated pieces, 7: watery) and gastrointestinal symptoms (excess flatulence in the rectum, abdominal distention, borborisms, abdominal pain and the occurrence of vomiting or nausea), will be assessed daily throughout the study period using a five-point scale (0: none, 1: weak, 2: moderate, 3: strong, 4: very strong).

In addition, the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire will be used to assess symptomatic evolution.

Before starting the intervention, each participant will record the frequency of defecation, characteristics and feeling of defecation (as an initial assessment) and daily after the start of the intervention.

They will fill out a questionnaire about bowel function weekly.

Changes in quality of life during the study will be measured by the SF-36 questionnaire, which consists of 36 items encompassed in 8 scales or components: functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects, mental health and another question of comparative evaluation between the current health conditions and that of a year ago.

The data will be organized and recorded in a database in the Microsoft Office Excel 2007® program with double entry. The statistical analysis will be performed in the Statistical statistical program Package for the Social Sciences (SPSS) version 24.0 for Windows.

Quantitative variables will be described and presented in mean and standard deviation from the mean if the distribution is symmetrical or in median and interquartile range if it is asymmetric. Nominal variables will be described in frequency categories as of the appearance in the described groups. To assess the distribution of data, the Shapiro-Wilk normality test will be applied. If the data is asymmetric, it will undergo logarithmic normalization or the non-parametric test will be used.

The intragroup changes will be analyzed by the difference (Basal and End) between the variables, using the paired Student t test or Wilcoxon.

When including 60% of patients, the data will be evaluated by an independent researcher to check whether the difference estimates are true. If necessary, the sample calculation will be reassessed

The assessment of treatment adherence will be measured by self-report on the daily assessment and telephone interviews, and at the end of the study you will be asked to deliver the supplement package.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes;
* Aged between 18 and 65 years;
* 24 hours after starting antibiotic treatment;
* Antibiotics tretament for a minimum of 3 days and a maximum of 14 days;
* Informed consent must be signed before starting the study.

Exclusion Criteria:

* blood pressure is outside the normal range (systolic blood pressure> 140, systolic blood pressure <90, diastolic> 90);
* history of heart disease, including heart valve disease or heart surgery, any implantable device;
* continuous or recent use of antibiotic therapy in the 30 days prior to the first administration of the study supplement;
* ostomates or users of parenteral nutrition;
* immunosuppressive therapy or any health condition that causes immunosuppression (including hematology malignancies, AIDS);
* Crohn's disease or ulcerative colitis;
* previous infection with Clostridium difficile documented less than 3 months before the start of the study;
* history of daily consumption of probiotics, fermented milk;
* individuals known to have demonstrated a previous reaction, including anaphylaxis, to any substance in the study product composition;
* individuals with active diarrhea (3 or more liquid stools per 24 hour period);
* pregnant women at the time of recruitment or planning to become pregnant during the study;
* Individuals with concomitant participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Decreased diarrhea | 10 - 14 days
  Decreased diarrhea through bristol scale. The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories. Categories: 1 - 7

SECONDARY OUTCOMES:
Improve in Quality of life | 10-14 days
  Improved quality of life through Short Form 36 Health Survey (SF-36) scale/questionare. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Improve of gastrointestinal symptoms | 10 - 14 days
  Improve of gastrointestinal symptoms through Gastrointestinal Symptom Rating Scale (GSRS). The GSRS is a disease-specific instrument. The 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Each item is rated on a 7-point Likert scale. Scale 7 refers to worse symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- GABBIA Biotecnologia, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided